CLINICAL TRIAL: NCT00478166
Title: Posterior Cingulate Function in Persons With Risk Factors for Alzheimer's Disease
Acronym: PC
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2004-174
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2011-04

CONDITIONS: Magnetic Resonance Imaging; Alzheimer's Disease; Dementia; Adult Children; Risk
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to use fMRI techniques to explore a certain part of the brain associated with Alzheimer's disease known as the posterior cingulate. Determining the functionality of this brain region may help us diagnose AD more accurately, thus allowing earlier treatment.

DETAILED DESCRIPTION:
The posterior cingulate is a key brain region suggested by recent studies to be affected in people at risk for Alzheimer's Disease (AD). Because the PC is affected very early in the course of AD and the region may have reduced function even prior to the onset of symptoms, further understanding of its functional role and its relationship to other brain regions may be helpful in detecting AD earlier and in monitoring disease progression and treatment. This project examines the role of the PC and its connections to other brain regions using functional magnetic resonance imaging (fMRI), a technique that allows us to examine the brain at work during tests of memory and decision-making. The main goal is to see if functional connections between brain regions are modulated by risk for AD.

ELIGIBILITY:
Inclusion Criteria:

* Cognitively healthy
* (Controls Only) Parents survived past age 70 and did/do not have memory problems.

Exclusion Criteria:

* Claustrophobia
* Metallic or electronic implants

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People who are enrolled in the Wisconsin Registry for AD Prevention (WRAP), recruited from Memory clinics and the community.
Sampling Method: Non-Probability Sample
Enrollment: 206 (Estimated)
Dates: Start 2005-07; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sterling C Johnson, PhD, Principal Investigator — University of Wisconsin/VA GRECC
Locations (1):
- University of Wisconsin - Wisconsin Comprehensive Memory Program, Madison, Wisconsin, United States

REFERENCES:
- See also: Johnson Imaging Lab website — http://www.brainmap.wisc.edu